CLINICAL TRIAL: NCT02463851
Title: PVAC GOLD Versus Irrigated RF Single Tip Catheter With Contact FORCE Ablation of the Pulmonary Veins for Treatment of Drug Refractory Symptomatic Paroxysmal and Persistent Atrial Fibrillation
Acronym: GOLD-FORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L.V.A. Boersma (Other)
Responsible Party: Sponsor-Investigator, L.V.A. Boersma, Cardiologist, R&D Cardiologie
Organization: R&D Cardiologie (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDC-2014.01
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: Ablation; Multi-electrode catheter PVAC; Single-tip catheter Contact Force; Holter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF-Ablation with Multi-electrode catheter (Active Comparator): Regular AF-ablation with a multi-electrode ablation catheter
  Interventions: Device: PVAC GOLD multielectrode catheter
- AF-Ablation with Contact Force single-tip electrode (Active Comparator): Regular AF-ablation with a regular Contact Force single-tip ablation catheter
  Interventions: Device: Contact Force single-tip ablation catheter

INTERVENTIONS:
Device: PVAC GOLD multielectrode catheter — Cardiac ablation for Atrial Fibrillation
  Arms: AF-Ablation with Multi-electrode catheter
Device: Contact Force single-tip ablation catheter
  Arms: AF-Ablation with Contact Force single-tip electrode

SUMMARY:
The GOLD FORCE trial investigates the differences between treatment with a Contact Force single-tip catheter against the PVAC GOLD multielectrode catheter in cardiac ablation procedures in patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. History of symptomatic paroxysmal atrial fibrillation defined as:

   * Self-terminating AF with episodes lasting no more than seven consecutive days before spontaneous conversion back to sinus rhythm
   * Documentation of one or more events with PAF tracings by ECG, event recordings, pacemaker strips or monitor rhythm strips within the past year
   * AF symptoms defined as the manifestation of any of the following:

     * Palpitations
     * Fatigue
     * Exertional dyspnea
     * Effort intolerance
2. Age between 18 and 70 Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study

Exclusion Criteria:

1. Structural heart disease of clinical significance including:

   * Previous cardiac surgery (excluding CABG)
   * Symptoms of congestive heart failure including, but not limited to, NYHA Class III or IV CHF and/or documented ejection fraction < 40% measured by acceptable cardiac testing
   * Left atrial diameter of > 45mm as measured in the parasternal long axis on transthoracic echocardiogram
   * LA volume>40 ml/m2
   * Stable/unstable angina or ongoing myocardial ischemia
   * Myocardial infarction (MI) within three months of enrollment
   * Aortic or mitral valve disease > Grade II
   * Congenital heart disease (not including ASD or PFO without a right to left shunt) where the underlying abnormality increases the risk of an ablative procedure
   * Prior ASD or PFO closure with a device using a percutaneous approach
   * Hypertrophic cardiomyopathy (LV wall thickness > 1.5 cm)
   * Pulmonary hypertension (mean or systolic PA pressure >50mm Hg on Doppler echo
2. Prior ablation for arrhythmias other than AF within the past three months
3. Prior left sided AF ablation
4. Enrollment in any other ongoing arrhythmia study protocol Any ventricular tachy-arrhythmias currently being treated where the arrhythmia or the management may interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2015-06; Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants free of Atrial Fibrillation and not taking anti-arrhythmic drugs | Month 3 after intervention

CONTACTS AND LOCATIONS:
Locations (3):
- Praxisklinik Herz und Gefäße, Dresden, Germany
- Netherlands (2):
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein, Utrecht
  - Isala Klinieken, Zwolle